CLINICAL TRIAL: NCT03882983
Title: A Phase I Safety Study Using Stromal Vascular Fraction From Lipoaspirate in the Treatment of Chronic Non-healing Wounds
Brief Title: Stromal Vascular Fraction From Lipoaspirate to Treatment of Chronic Non-healing Wound
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Antria (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CW0001
Record Dates: First submitted 2017-05-24; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Chronic Wounds
Keywords: Autologous Adult Stem Cell; Lipoaspirate; Non-healing Wounds; Stomal Vasular Fraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antria Cell Preparation Process (Experimental): Safety will be evaluated by collection of vital signs, EKG, patient surveys, and assessments
  Interventions: Drug: Antria Cell Preparation Process

INTERVENTIONS:
Drug: Antria Cell Preparation Process — Biological/Vaccine: Stromal Vascular Fraction The SVF obtained from adipose tissue will be added to the graft
  Other Names:
  * Stromal Vascular Fraction
  * Adiployx Biological/Vaccine:
  Other Names: SVF

SUMMARY:
This is a Phase I, open-label, single arm study to demonstrate the safety of Antria Cell Preparation Process during fat grafting augmented with autologous adipose derived stromal vascular fraction to demonstrate the safety and efficacy of administration of SVF enriched fat grafting in chronic wounds

DETAILED DESCRIPTION:
This is a Phase I, open-label, single arm study to demonstrate the safety of Antria Cell Preparation Process during fat grafting augmented with autologous adipose derived stromal vascular fraction to demonstrate the safety and efficacy of administration of SVF enriched fat grafting in chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male, Age 18 years or older
2. Subjects that are diagnosed with one or more chronic wounds.
3. Able to understand and provide written and verbal informed consent

Exclusion Criteria:

1. Currently taking or have taken NSAIDs within last two weeks or corticosteroids within the last six weeks prior to screening.
2. Diagnosis of any of the following medical conditions:

   * Active malignancy (diagnosed within 5 years), except for treated non-melanoma skin cancer or other non-invasive or in-situ neoplasm (e.g. cervical cancer)
   * Active infection (other than their wound)
3. Subjects who are unlikely to comply with the protocol (e.g., uncooperative attitude, inability to return for subsequent visits, dementia, and/or otherwise considered by the Investigator to be unlikely to complete the study)
4. Subjects with a known drug or alcohol dependence within the past 12 months as judged by the Investigator
5. Any other disease condition or laboratory results that in the opinion of the investigator may be clinically significant and render the subject inappropriate for the study procedure(s), may alter the accuracy of study results, or increase the risk for subjects.
6. Subjects with life-expectancies less than 12 months
7. Subjects with known collagenase allergies
8. Pregnant females On radiotherapy or chemotherapy agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Bates-Jensen Wound Assessment | 1 year
  This assessment focuses on analysis wounds with regards to the following information: size, depth, edges, undermining, necrotic tissue type, necrotic tissue amount, exudate type, exudate amount, skin color surrounding the wound, peripheral tissue edema and induration, granulation tissue, and epithelialization. Each item will be measured on a scale 1-5. A score of 1 will indicate least severe and a score of 5 will indicate the most severe.

SECONDARY OUTCOMES:
Digital Picture of wound | 1 year
  Digital pictures of subject's wounds pre-treatment and post-treatment will be performed to show changed from baseline assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E Maliver, MD, Principal Investigator — Antria Inc.
Locations (1):
- Indiana Regional Medical Center, Indiana, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No